CLINICAL TRIAL: NCT06274229
Title: Anonymous Survey Among Local Residents on the Impact of the Planned Measures in the Five Partner Cities of the DivAirCity Project on Their Social Life, Health and Well-being
Brief Title: DivAirCity Social Health Survey
Acronym: DivAirCitySH
Status: Recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universitat Politècnica de València (Other); Universitatea din Bucuresti (Other); University of Aarhus (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); European Commission (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr., Charite University, Berlin, Germany
Other Study IDs: EA4/252/23
Record Dates: First submitted 2024-02-02; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Psychological Stress; Psychological Well-Being; Pollution; Exposure
Keywords: Traffic noise; Air pollution; General Health condition
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being | interventions — Air Pollution

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Aarhus, installation site: Residents of Aarhus (DK), living at or nearby the site of the installed Intervention
  Interventions: Other: Air pollution and noise reducing installations
- Aarhus, control site: Residents of Aarhus (DK), living at or nearby the control site
- Bucharest, intervention site: Residents of Bucharest (RO), living at or nearby the site of the installed Intervention
  Interventions: Other: Air pollution and noise reducing installations
- Bucharest, control site: Residents of Bucharest (RO), living at or nearby the control site
- Castelló, intervention site: Residents of Castelló (ES), living at or nearby the site of the installed Intervention
  Interventions: Other: Air pollution and noise reducing installations
- Castelló, control site: Residents of Castelló (ES), living at or nearby the control site
- Orvieto, intervention site: Residents of Orvieto (IT), living at or nearby the site of the installed Intervention
  Interventions: Other: Air pollution and noise reducing installations
- Orvieto, control site: Residents of Orvieto (IT), living at or nearby the control site
- Potsdam, intervention site: Residents of Potsdam (DE), living at or nearby the site of the installed Intervention
  Interventions: Other: Air pollution and noise reducing installations
- Potsdam, control site: Residents of Potsdam (DE), living at or nearby the control site

INTERVENTIONS:
Other: Air pollution and noise reducing installations — A number of means to reduce traffic noise and traffic exhausts and improve air quality will be implemented at designated urban spaces (intervention sites), while other places with comparable amount of traffic and no such changes will serve as control sites.
  Groups: Aarhus, installation site; Bucharest, intervention site; Castelló, intervention site; Orvieto, intervention site; Potsdam, intervention site

SUMMARY:
To reduce stress among urban residents, the consortium members of the European Council Horizon 2020 research program DivAirCity install different stress reducing, noise reducing and air quality improving means in the five cities of the consortium. This study measures physiological and psychological stress and health factors before and after the implementation of the project (at intervention sites) and compares the change (improvement) to the change in comparable places where no means were installed (control site).

DETAILED DESCRIPTION:
Scientific studies show that increased stress can favor the development of e.g. high blood pressure, heart disease, mental illness, infectious diseases, headaches and sleep disorders. This means that stress causes considerable costs for western healthcare systems, including in our city and this neighbourhood. In large cities, where there are often hardly any natural green and forest areas left, depression and anxiety syndromes, for example, are more common than among the rural population.

For example, in Germany, more than three quarters of the population live in densely or moderately populated areas, while the global average is more than 50 per cent. Due to increasing urbanisation, people living in cities will be heavily dependent on urban nature, which can be a relevant health-promoting factor. Several studies have shown that natural spaces such as city parks, parks and even greenery on streets have a positive impact on the health of residents, both individually and collectively.

The European Council Horizon 2020 project DivAirCity (acronym explanation in the text below) is about making formerly busy public spaces in European cities more attractive again for residents and citizens. The aim is to redesign the spaces in such a way that people of different age groups, social classes and identities ("Div") can (once again) come together and meet in these places on a daily basis. To this end, these places are to be changed through various installations (planting trees, redesigning parks, shading, watering in summer) in such a way that the local air quality ("Air") in the cities ("City") improves significantly. This is realized on the one hand by installing air quality measuring equipment and by recording the number of people and the time they spend in these places (objective measurements).

In addition to these objective measurements, this study records the impact on psychological and physiological health that the installations (intervention) has on the residents. To this end, it will be measured how residents feel in terms of quality of life, current stress, general health, and whether they feel safe and secure in the specific place (comfort, safety and security) and whether they enjoy going there and staying there,. These measurements will take place both before (day -60 to day -30) and after (day +30 and day +60) the installment of the intervention.

Finally, we would like to know your age group, your gender and how close you live to the location of the conversion/installation. We would like to invite you to take part in this survey again after the remodelling project.

ELIGIBILITY:
Inclusion Criteria:

* Participants must live or work at or near the installation (intervention group) or control site (control group)

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of the five cities (18+ years of age)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
WHO-5 Well-being Scale | Baseline: 60 to 30 days before the installation implementation vs Posttest: 30 to 60 days after the installation has been implemented
  Validated Questionnaire

SECONDARY OUTCOMES:
Kessler K6 psychological distress | Baseline: 60 to 30 days before the installation implementation vs Posttest: 30 to 60 days after the installation has been implemented
  Validated Questionnaire
ASKU questionnaire | Baseline: 60 to 30 days before the installation implementation vs Posttest: 30 to 60 days after the installation has been implemented
  Validates Questionnaire for self-efficacy

OTHER OUTCOMES:
Questionnaire for General Physiological Health | Baseline: 60 to 30 days before the installation implementation vs Posttest: 30 to 60 days after the installation has been implemented
  Custom-made Questionnaire
Questionnaire about feelings of safety and security at the site | Baseline: 60 to 30 days before the installation implementation vs Posttest: 30 to 60 days after the installation has been implemented
  Custom-made Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof MD, Principal Investigator — Charite Universitaetsmedizin Berlin
Locations (1):
- Charité -- Universitaetsmedizin Berlin, Berlin, Germany